CLINICAL TRIAL: NCT05476263
Title: Non-interventional, Observational, Prospective, Multicentre Study in a Routine Clinical Care Setting Using a Marketed Medical Device in Line With the Corresponding IFU in the Intended Patient Population
Brief Title: Suprasorb® CNPendo Used for Negative Pressure Therapy in the Oesophagus and Rectum to Support Defect and Wound Healing
Acronym: Velox
Status: Recruiting | Type: Observational
Sponsor: Lohmann & Rauscher (Industry)
Collaborators: CRI-The Clinical Research Institute GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-03
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2024-09

CONDITIONS: Esophagus Injury; Rectal Lesion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A Post-Market Clinical Follow-up (PMCF) study designed as non-interventional, observational, prospective, multicentre study in a routine clinical care setting using a marketed medical device in line with the corresponding Instruction for Use (IFU) in the intended patient population.

Patients will be diagnosed and evaluated for eligibility in routine clinical care by expert centres in the indication of interest. They will be consecutively enrolled into the study provided that all inclusion and exclusion criteria are met and written consent is given to use their clinical routine data according to data privacy regulations.

The study protocol does not define specific study procedures for patients enrolled. Therapies and procedures during the course of this study will be performed according to the decision of the treating physician based on current applicable medical guidelines and on local policy in clinical routine care.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Acute transmural defects, injuries and wounds in oesophagus or rectum, including perforations (iatrogenic or spontaneous) and anastomotic insufficiencies (Index defect)
* Indication of treatment with Suprasorb® CNPendo system according to IFU and medical guidelines
* Signed informed consent for usage of data

Exclusion Criteria:

* Pre-existing coagulation disorders with increased risk of bleeding
* Defects involving the bronchial system (bronchus/trachea/pulmo)
* Any foreseeable deviation from IFU of Suprasorb® CNP endo
* Known intolerance or allergy to one or more components of Suprasorb® CNPendo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female and male patients with acute defects, injuries and wounds in the oesophagus or rectum and an indication of treatment with Suprasorb® CNPendo system according to IFU and medical guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Time period in days from index use of Suprasorb® CNPendo to release for oral food intake (in upper GI tract use) or release for stoma relocation (in lower GI tract use). | 3 months
  Time period in days from index use of Suprasorb® CNPendo to release for oral food intake (in upper GI tract use) or release for stoma relocation (in lower GI tract use).
  In case of lower GI tract use and no stoma present, time period to release for oral food intake is the relevant endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Laukötter, Prof., MD, Principal Investigator — Klinikum Rheine, Mathias-Spital
Locations (7):
- Germany (7):
  - Uniklinik Berlin Charite, Berlin
  - Central Interdisciplinary Endoscopy, II. Medical Clinic Mannheim Medical University, Mannheim
  - Clinic for general, visceral and transplant surgery at the University of Munich, Munich
  - Uniklinik MRI, Munich
  - Universitätsklinikum Münster (UKM) Klinik für Allgemein-, Viszeral- und Transplantationschirurgie, Münster
  - Klinikum Rheine, Mathias-Spital, Chirurgische Klinik I: Allgemein- und Viszeralchirurgie, Rheine
  - Universitätsklinikum Tübingen, Innere Medizin I - Gastroenterologie, Gastrointestinale Onkologie, Hepatologie, Infektiologie und Geriatrie, Tübingen

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT05476263/Prot_000.pdf